CLINICAL TRIAL: NCT06054724
Title: Comparison of Yoga-Based and Pilates-Based Respiratory Training Effect for Individuals with Urinary Incontinence
Brief Title: Yoga and Pilates Based Respiratory Training Effect for Individuals with Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Şevval Zeynep Girit, Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulUCSZG
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-05

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; yoga; pilates; respiratory training
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga-based Respiration Group (Experimental): This group will be given yoga-based breathing exercises
  Interventions: Other: Yoga-Based Respiration Training
- Pilates-based Respiration Group (Experimental): This group will be given pilates-based breathing exercises
  Interventions: Other: Pilates-Based Respiration Training

INTERVENTIONS:
Other: Yoga-Based Respiration Training — The selected asanas, believed to be beneficial for urinary incontinence, will be practiced with a focus on breath. After the assessment session, participants will engage in three days of face-to-face yoga sessions. On the days when face-to-face sessions are held, participants will perform the second session on their own at home. The exercises will be progressively intensified during the 3rd and 5th weeks to ensure progression. The exercise program will be conducted at home, with approximately 20-minute sessions, twice a day, five days a week, for a total of 6 weeks.
  Arms: Yoga-based Respiration Group
Other: Pilates-Based Respiration Training — Before starting the 6-week practice protocol, participants will be taught the transversus abdominis muscle activation and centering, pilates-specific lateral costal breathing and other key elements of pilates. Pilates exercises chosen as beneficial for urinary incontinence will be performed with a focus on breath. After the assessment session, participants will engage in three days of face-to-face pilates sessions. On the days when face-to-face sessions are held, participants will perform the second session on their own at home. The exercises will be progressively intensified during the 3rd and 5th weeks to ensure progression. The exercise program will be conducted at home, with approximately 20-minute sessions, twice a day, five days a week, for a total of 6 weeks.
  Arms: Pilates-based Respiration Group

SUMMARY:
The aim of the study is to examine and compare the effects of yoga-based and pilates-based respiratory training on incontinence severity, pelvic floor muscle function and quality of life in the rehabilitation of individuals with urinary incontinence.

DETAILED DESCRIPTION:
In the literature, it has been stated that the pelvic floor alone does not play a singular role in maintaining continence, but rather forms a functional unit with the diaphragm, abdominal, and spinal muscles. Since the inability of any of these structures to perform their function properly negatively affects the function of the others, normalization and optimal functioning of the pelvic floor-thoracic diaphragm relationship are crucial in individuals with urinary incontinence. This study aims to investigate the effectiveness of yoga and Pilates approaches, considering breath as a fundamental building block, through respiration-based training programs in women with urinary incontinence.

The participants who volunteered to take part in the study will be randomly divided into two groups, namely the Yoga-based Respiration Group (Group 1) and the Pilates-based Respiration Group (Group 2), using a computer-assisted randomization program. After the groups are assigned, the initial three sessions for both groups will be conducted face-to-face under the guidance of a physiotherapist to ensure the correct execution of the exercises. The exercise program for both groups will consist of approximately 20-minute sessions, with two sessions per day, five days a week, for a total of six weeks. On the days when face-to-face sessions are held, one session will be conducted in-person, while the other session will be performed at home. During the 3rd and 5th weeks, the exercises will be progressively intensified for both groups to ensure progression, and patients will be called for face-to-face sessions. At the end of the six weeks, patients will undergo face-to-face evaluations once again.

ELIGIBILITY:
Inclusion Criteria:

* Having the diagnosis of stress or mixed urinary incontinence.
* Being volunteer to participate in the study.
* Having planned routine treatment program and being compliant with treatment
* Having no obstacles for the planned assessments.
* People who capable of written, verbal and visual communication

Exclusion Criteria:

* Having received treatment for urinary incontinence in the last 3 months.
* Using medication for vaginal or urinary tract infections.
* Pregnancy.
* Being within the first 3 years postpartum.
* Presence of concurrent pulmonary, neurological, rheumatological, or musculoskeletal disorders affecting spinal alignment.
* History of surgery that may impede the exercise planned within the scope of the study.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 46 (Actual)
Dates: Start 2023-08-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) | baseline and post-intervention (7th week)
  International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) is used to measure the severity of incontinence. This form includes questions about the frequency and amount of urinary incontinence, its effect on daily life and the causes of urinary incontinence, and an evaluation is made for the last 4 weeks. It is calculated by summing the scores of the 3 dimensions in the test, and a result in the range of 0-21 points is obtained.
24-Hour Pad Test | baseline and post-intervention (7th week)
  24-hour pad test The 24-Hour Pad Test is an objective evaluation method used to determine the severity of urinary incontinence. Patients are asked to start the test with an empty bladder. It is requested that the used pad should be changed every 4-6 hours and kept in a locked bag until it is taken to the hospital. Patients use the same type of pad throughout the test and are asked to bring an unused pad of the same type when coming to the hospital. The amount of urinary incontinence is calculated by subtracting the weight of the clean pad from the weight of the pads accumulated within 24 hours. It is classified as 4-20 g mild, 21-74 g moderate, >75 g severe urinary incontinence.
PFM Function- MyoPlusPro EMG Device | baseline and post-intervention (7th week)
  Pelvic floor muscle function will be evaluated with electromyographic measurement (EMG). Before the test, participants will be asked to empty their bladders and will be taught to contract and relax the isolated pelvic floor muscle. Surface active electrodes will be placed to the right and left of the perineal body, and they will be asked to make 5 maximal contractions and 5 relaxations, and the obtained values will be recorded in μV.
Incontinence Quality of Life Questionnaire (I-QOL) | baseline and post-intervention (7th week)
  Incontinence Quality of Life Questionnaire (I-QOL) includes questions that examine limitation of behavior, psychosocial influence and social isolation. Questions are scored between 1 and 5, and high scores indicate good quality of life.
Incontinence Impact Questionnaire Short Form (IIQ-7) | baseline and post-intervention (7th week)
  The Incontinence Impact Questionnaire (IIQ-7) is used to measure the impact of urinary incontinence on individuals' daily and social lives and participation. The survey contains 7 questions, each question is scored between 1 and 4. High scores indicate negative impact.

SECONDARY OUTCOMES:
Core Muscle Endurance Assessment | baseline and post-intervention (7th week)
  The endurance of the core muscles will be evaluated with the McGill Core Endurance Test Battery. The test has 4 stages; Trunk Flexor Endurance Test Lateral Flexor Endurance Test Trunk Extensor Endurance Test
Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) assessment | baseline and post-intervention (7th week)
  Maximum inspiratory pressure (MIB) and maximum expiratory pressure (MEP) measurements will be made to assess respiratory function. During the MIB measurement, the participant is asked to make a maximal expiration and maximally inhale at the end of the expiration, and during the MEP measurement, to make a maximal inspiration and then a maximal expiration. Each measurement is repeated 3 times and the best value is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sevval Z Girit, Principal Investigator — Istanbul University - Cerrahpasa; Ipek Yeldan, Prof., Study Chair — Istanbul University - Cerrahpasa
Locations (2):
- Turkey (Türkiye) (2):
  - Basaksehir Cam ve Sakura City Hospital, Istanbul, Basaksehir
  - Istanbul University-Cerrahpasa, Istanbul, Buyukcekmece

IPD SHARING:
Plan to Share IPD: No